CLINICAL TRIAL: NCT01252680
Title: A Randomized, Double-blind Clinical Trial of Two Inactivated Hepatitis A Vaccines in Healthy Children
Brief Title: Immunogenicity and Interchangeability of Two Inactivated Hepatitis A Vaccines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: PRO-HA-4014
Record Dates: First submitted 2010-11-29; First posted 2010-12-03 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Hepatitis A
MeSH Terms: conditions — Hepatitis A | interventions — Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: Healive+Healive (Experimental): 75 subjects to receive two doses of Healive 6 months apart
  Interventions: Biological: Healive+Healive
- Group 2: Healive+Havrix (Experimental): 75 subjects to receive one dose of Healive and another dose of Havrix 6 months apart
  Interventions: Biological: Healive+Havrix
- Group 3: Havrix+Havrix (Experimental): 75 subjects to receive two doses of Havrix 6 months apart
  Interventions: Biological: Havrix+Havrix
- Group 4: Havrix+Healive (Experimental): 75 subjects to receive one dose of Havrix and another dose of Healive 6 months apart
  Interventions: Biological: Havrix+Healive

INTERVENTIONS:
Biological: Healive+Healive — Hepatitis A vaccine (Healive), 250 u per dose per 0.5 millilitre. Vaccines will be administered two doses in the deltoid muscle of the arm 6 months apart
  Other Names: Hepatitis A vaccine
  Arms: Group 1: Healive+Healive
Biological: Healive+Havrix — Two kinds of Hepatitis A vaccines, Healive(250 u per dose per 0.5 millilitre) and Havrix(720 ELU per dose per 0.5 millilitre). The first dose will be administered with Healive, followed by another dose of Havrix after 6 months
  Other Names: Hepatitis A vaccine
  Arms: Group 2: Healive+Havrix
Biological: Havrix+Havrix — Hepatitis A vaccine (Havrix), 720 ELU per dose per 0.5 millilitre. Vaccines will be administered two doses in the deltoid muscle of the arm 6 months apart
  Other Names: Hepatitis A vaccine
  Arms: Group 3: Havrix+Havrix
Biological: Havrix+Healive — Two kinds of Hepatitis A vaccines, Healive(250 u per dose per 0.5 millilitre) and Havrix(720 ELU per dose per 0.5 millilitre). The first dose will be administered with Havrix, followed by another dose of Healive after 6 months
  Other Names: Hepatitis A vaccine
  Arms: Group 4: Havrix+Healive

SUMMARY:
This is a randomized, double-blind clinical trial of two inactivated hepatitis A vaccines in healthy children, immunogenicity and interchangeability of the two inactivated hepatitis A vaccines were evaluated.

DETAILED DESCRIPTION:
This was a monocenter, comparative trial in which healthy children were randomized to receive two doses of hepatitis A vaccine 6 months apart. The trial was conducted in accordance with the Edinburgh version of the Declaration of Helsinki. The study was approved by the Ethics Committee. Parents or legal guardians of all participants gave written informed consent prior to study entry. Eligible subjects were between 18m and 6 years of age, When enrolled, children were randomized to four equal groups with different intervention. Immunogenicity and interchangeability of two inactivated hepatitis A vaccines were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged between 1.5 and 5 years, with no history of hepatitis A virus infection or hepatitis A vaccine vaccination
* Provided birth certification or vaccination card
* Parent(s) or legal guardian(s) are able to understand and sign the informed consent

Exclusion Criteria:

* Axillary temperature > 37.0 centigrade at the time of dosing
* Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine
* Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
* Autoimmune disease or immunodeficiency
* Congenital malformation, developmental disorders or serious chronic diseases (such as Down's syndrome, diabetes, sickle cell anemia or neurological disorders)
* Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
* History or family history of convulsions, epilepsy, brain disease and psychiatric
* History of any blood products within 3 months
* Administration of any other investigational research agents within 30 days
* Administration of any live attenuated vaccine within 30 days
* Administration of subunit or inactivated vaccines within 14 days
* Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent

Ages: 18 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 303 (Actual)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Immunogenicity and interchangeability of two inactivated hepatitis A vaccines | 7 months

SECONDARY OUTCOMES:
safety of two inactivated hepatitis A vaccines | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-lun Zhang, Principal Investigator — Tianjin Centers for Diseases Control and Prevention
Locations (1):
- Tianjin Centers for Diseases Control and Prevention, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Zhang ZL, Zhu XJ, Wang X, Liang M, Sun J, Liu Y, Gao ZG, Wu JY, Dong XJ, Liu RK, Chen JT, Zhang YQ, Wang W, Zhang LP, Yin W. Interchangeability and tolerability of two inactivated hepatitis A vaccines in Chinese children. Vaccine. 2012 Jun 8;30(27):4028-33. doi: 10.1016/j.vaccine.2012.04.038. Epub 2012 Apr 23. PMID 22537990